CLINICAL TRIAL: NCT00490737
Title: An Evaluation of the Pharmacokinetic Profile and Safety and Tolerability of Multiple Doses of 6mg/kg Intravenous Daptomycin in Non-Infected Adult Subjects With End Stage Renal Disease on Hemodialysis or Continuous Ambulatory Peritoneal Dialysis
Brief Title: Safety Study to Evaluate Daptomycin in Non-infected Adults Who Are Either on Hemodialysis or Continuous Ambulatory Peritoneal Dialysis (MK-3009-021)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3009-021; DAP-REN-07-01 (Other: Cubist Study Number)
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: End-Stage Renal Disease
Keywords: ESRD; dialysis; hemodialysis; continuous ambulatory peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hemodialysis (HD) Participants (Experimental): Participants will receive daptomycin 6 mg/kg by intravenous infusion (i.v.) at 48-hours intervals (with dialysis) for a total of 3 doses.
  Interventions: Drug: daptomycin
- Continuous Ambulatory Peritoneal Dialysis (CAPD) Participants (Experimental): Participants will receive daptomycin 6 mg/kg, i.v., at 48-hours intervals for a total of 3 doses.
  Interventions: Drug: daptomycin

INTERVENTIONS:
Drug: daptomycin — 6mg/kg, i.v. infusion over 30 minutes; every 48 hours for a total of 3 doses
  Other Names: Cubicin

SUMMARY:
This study is to examine the safety of daptomycin in patients with End Stage Renal Disease.

DETAILED DESCRIPTION:
This is an open label, non-randomized, non-comparative Phase 1 study designed to evaluate the PK profile, safety and tolerability of intravenous ( i.v.) daptomycin. Non-infected subjects with end stage renal disease undergoing hemodialysis (HD) or continuous ambulatory peritoneal dialysis (CAPD) will be enrolled in this in-patient study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study-related procedure not part of normal medical care;
* Considered to be in appropriate health for study entry by the Investigator (e.g., no acute, debilitating medical problems) and appropriate candidate for completing study treatment;
* Male or female >18 years of age;
* If female of childbearing potential; willing to practice reliable birth control measures during study treatment, not lactating/pregnant, has a documented negative pregnancy test result within 24 hours prior to study medication administration, and willing to practice effective means of birth control for >28 days after study completion;
* If taking concomitant medications, subject must be on a relatively stable dose for at least two weeks prior to study medication administration;
* Functioning dialysis access (e.g. graft or fistula) for subjects undergoing HD and functioning dialysis access (e.g. peritoneal catheter) for subjects undergoing CAPD;
* ESRD on stable HD regimen of thrice weekly sessions with high-flux membranes or stable CAPD regimen.

Exclusion Criteria:

* If female, pregnant or lactating;
* Received an investigational drug (including experimental biologic agents) within 30 days of study entry;
* Evidence of active ongoing infection;
* Unable to discontinue use of HMG-CoA reductase inhibitor therapy for duration of study;
* Has received any dose(s) of daptomycin within 5 days prior to receiving the first dose of study drug;
* Known to be allergic or intolerant to daptomycin;
* Body Mass Index (BMI) < 18.5 or > 40 kg/m2 [BMI = weight (kg)/height (m2)];
* WBC >12, 000 cells/mm3 or <2500 cells/ mm3;
* Baseline creatinine phosphokinase (CPK) values >3X ULN (upper limit of normal);
* Alanine aminotransferase (ALT) >5X ULN;
* Aspartate aminotransferase (AST) >5X ULN;
* Known HIV-infected subjects with CD4 count ≤200 cells/mm3;
* Hemoglobin < 9 gm/dL;
* Active illicit drug and/or alcohol abuse;
* Myocardial infarction within last 6 months;
* Hospitalized for non-vascular or peritoneal dialysis (PD) access issues within 30 days;
* Subjects with a history of muscular disease (e.g., polymyositis, muscular dystrophy);
* Subjects with a history of neurological disease (e.g., Guillain Barré, multiple sclerosis), except stroke >6 months prior to study entry;
* Intramuscular injection within 7 days of study drug administration;
* Has a moribund clinical condition (i.e., high likelihood of death during the next 3 days);
* Is considered unlikely to comply with study procedures or to return for scheduled post-treatment evaluations;
* Neutropenic subjects with absolute neutrophil count ≤500 cells/mm3 History of rhabdomyolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08-12 (Actual); Primary Completion 2008-05-12 (Actual); Study Completion 2008-05-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Study Day 1, 3, 5 and 7 or 8

SECONDARY OUTCOMES:
Safety and Tolerability | Study Days 1 through 16 or 17

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Benziger DP, Pertel PE, Donovan J, Yankelev S, Schwab RJ, Swan SK, Cannon C. Pharmacokinetics and safety of multiple doses of daptomycin 6 mg/kg in noninfected adults undergoing hemodialysis or continuous ambulatory peritoneal dialysis. Clin Nephrol. 2011 Jan;75(1):63-9. PMID 21176752